CLINICAL TRIAL: NCT03667794
Title: Evaluation of Novel Lung Function Parameters in Patients With Pulmonary Hypertension (PH)
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-PH
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Plethysmography, Whole Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PH patients: Patients with known or first diagnosis of PH
  Interventions: Diagnostic Test: body plethysmography; Diagnostic Test: impulse oscillometry; Diagnostic Test: multiple breath washout
- healthy controls: Healthy controls had normal lung function testing including whole-body plethysmography and transfer factor, no previously diagnosed pulmonary disease as well as no respiratory symptoms.
  Interventions: Diagnostic Test: body plethysmography; Diagnostic Test: impulse oscillometry; Diagnostic Test: multiple breath washout
- non-healthy controls: Non-healthy controls were allowed to have stable pulmonary comorbidities including chronic obstructive pulmonary disease (COPD), sarcoidosis, asthma, or fibrosis as well as non-pulmonary comorbidities.
  Interventions: Diagnostic Test: body plethysmography; Diagnostic Test: impulse oscillometry; Diagnostic Test: multiple breath washout

INTERVENTIONS:
Diagnostic Test: body plethysmography — measurement of conventional lung function parameters
Diagnostic Test: impulse oscillometry — measurement of central and peripheral airway resistance
Diagnostic Test: multiple breath washout — measurement of ventilation heterogeneity

SUMMARY:
Little is known about affection of small airways in patients with pulmonary hypertension as well as the ideal diagnostic approach. The investigators therefore aimed to evaluate novel or not widely used lung function tests for the evaluation of airway function in patients with PH.

ELIGIBILITY:
Inclusion Criteria:

* known or first diagnosis of PH

Exclusion Criteria:

* inability to perform lung function testing
* unable or unwilling to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PH group: known or first diagnosis of PH
  Healthy controls: normal lung function testing including whole-body plethysmography and transfer factor, no previously diagnosed pulmonary disease as well as no respiratory symptoms.
  Non-healthy controls: stable pulmonary comorbidities including COPD, sarcoidosis, asthma, or fibrosis as well as non-pulmonary comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
LCI | 30 minutes
  between-group difference in lung clearance index (LCI)
D5-20 | 30 minutes
  between-group difference in frequency dependence of resistance (D5-20)

SECONDARY OUTCOMES:
Discrimination small airway resistance | 30 minutes
  Evaluation of discriminative capability of impulse oscillometry
Discrimination ventilation heterogeneity | 30 minutes
  Evaluation of discriminative capability of multiple breath washout

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Trinkmann, MD, Principal Investigator — Universitätsmedizin Mannheim

IPD SHARING:
Plan to Share IPD: No